CLINICAL TRIAL: NCT01744171
Title: A Phase I Trial of a Recombinant Human hsp110-gp100 Chaperone Complex Vaccine for Advanced Stage IIIB/C or IV Melanoma
Brief Title: Vaccine Therapy in Treating Patients With Advanced Stage III-IV Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was Suspended since 2018; PI decided to terminate.
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 215912; NCI-2012-02231 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 215912 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Recurrent Melanoma; Stage IIIB Skin Melanoma; Stage IIIC Skin Melanoma; Stage IV Skin Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (recombinant hsp110-gp100 chaperone complex vaccine) (Experimental): Patients receive recombinant hsp110-gp100 chaperone complex vaccine ID on days 1, 15, and 43 in the absence of unacceptable toxicity.
  Interventions: Biological: Recombinant Human Hsp110-gp100 Chaperone Complex Vaccine; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Recombinant Human Hsp110-gp100 Chaperone Complex Vaccine — Given ID
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of vaccine therapy in treating patients with stage III-IV melanoma that has spread to other places in the body and usually cannot be cured or controlled with treatment (advanced). Vaccines made from peptides or antigens may help the body build an effective immune response to kill tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and clinically appropriate dose of human heat shock protein (hsp)110-gp100 chaperone complex melanoma vaccine (recombinant hsp110-gp100 chaperone complex vaccine) to recommend a phase II dose in stage IIIB/C and stage IV metastatic melanoma patients.

SECONDARY OBJECTIVES:

I. To examine the effect of the recombinant human hsp110-gp100 chaperone complex vaccine on measurable clinical tumor.

II. To determine gp100 and hsp110 specific cell mediated and humoral immune responses elicited by the chaperone complex vaccine.

III. To determine the effect of dose and serial administration of the chaperone complex vaccine on cell mediated and humoral immune responses.

IV. To quantify patient characteristics (human leukocyte antigen [HLA] subtype, immune cell function, etc.) that may correlate with immune response to the chaperone complex vaccine.

OUTLINE: This is a dose-escalation study.

Patients receive recombinant hsp110-gp100 chaperone complex vaccine intradermally (ID) on days 1, 15, and 43 in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Absolute neutrophil count (ANC) > 1500/uL
* Platelets >= 120,000/uL
* Total bilirubin =< 1.5 mg/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 1.5 x upper limit of normal (ULN)
* Serum creatinine =< 1.5 mg/dL (if > 1.5 mg/dL, then creatinine clearance should be > 60 mL/min)
* Blood urea nitrogen (BUN) =< 1.5 x ULN
* Have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria or physical exam
* An anticipated overall survival of at least 6 months
* Patients of child-bearing potential must agree to use acceptable contraceptive methods (e.g., double barrier) during treatment
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Patients must have undergone/undergo testing for v-raf murine sarcoma viral oncogene homolog B1 (BRAF) V600 mutation status
* Patients must have documented, clinically measurable 7th edition American Joint Committee on Cancer (AJCC) stage IIIB/C (bulky nodal and/or in transit disease) or stage IV (distant metastatic) melanoma; patients with brain metastases that have been appropriately treated with surgical resection and/or radiation are eligible for inclusion if they meet the performance status and life expectancy criteria; patients who are BRAF V600E mutation positive need to have failed, refused, or be ineligible for at least 2 lines of therapy (vemurafenib plus one other regimen)
* Stage IIIB/C patients must have refused, be ineligible for, or have failed at least one standard of care regional therapy (isolated limb perfusion or infusion) or one non-vaccine based systemic therapy (such as, high dose interleukin [IL]-2, dacarbazine/temozolomide, ipilimumab, or participation in a clinical trial); patients who are BRAF V600E mutation positive need to have failed, refused, or be ineligible for at least 2 lines of therapy (vemurafenib plus one other regimen)
* Stage IV patients must have refused, be ineligible for, or have failed at least one non-vaccine based systemic therapy (such as, high dose IL-2, dacarbazine/temozolomide, ipilimumab, or participation in a clinical trial); patients who are BRAF V600E mutation positive need to have failed, refused, or be ineligible for at least 2 lines of therapy (vemurafenib plus one other regimen)

Exclusion Criteria:

* Pregnant or nursing female patients
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the patient an unsuitable candidate to receive study drug
* Received an investigational agent within 30 days prior to enrollment
* Melanoma specific systemic therapy within 30 days of enrollment
* A history of AJCC stage IIIB/C or stage IV melanoma but no current clinical evidence of metastatic disease
* Known immunosuppressed conditions or active immunosuppressive therapy such as organ transplantation (including bone marrow transplant), high dose steroids, or human immunodeficiency virus (HIV); although a documented negative HIV test is not mandatory for enrollment, patients felt to have a high clinical suspicion for HIV will need to test negative prior to enrollment; use of topicals or eye drops containing steroids is acceptable; inhaled steroids are excluded
* Known autoimmune conditions including but not limited to rheumatoid arthritis, multiple sclerosis, lupus, scleroderma, sarcoidosis, vitiligo, inflammatory bowel disease, idiopathic thrombocytopenia purpura, Graves' disease, or Hashimoto's thyroiditis
* Previous history of splenectomy or whole spleen radiation
* Systemic immunoglobulin therapy within the last 30 days
* Previous history of anaphylaxis or severe allergic reaction to hsp110, gp100, other vaccines, or unknown allergens
* Previous or active non-melanoma malignancies (excluding non-melanoma skin cancer or carcinoma in situ of the cervix) diagnosed/treated within the last 5 years
* Active uncontrolled bacterial, viral, or fungal infection until these conditions are corrected or controlled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-03-26 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-06-11 (Actual)

PRIMARY OUTCOMES:
MTD of recombinant human hsp110-gp100 chaperone complex melanoma vaccine based on the probability of dose-limiting toxicity (DLT), graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4 | Up to 30 days after the last vaccine dose
  DLT is defined as grade 3 or 4 toxicity or grade 3 injection site toxicity, with the exception of grade 3 rigors/chills which will be tolerated for 48-72 hours if attributable to vaccine reaction.

SECONDARY OUTCOMES:
Objective tumor response according to RECIST version 1.1 | Up to 6 months
  Recombinant hsp110-gp100 chaperone complex vaccine specific cell mediated and humoral immune responses elicited by the chaperone complex vaccine as well as the effect of dose and serial administration on these responses will be assessed through the correlative science studies.

CONTACTS AND LOCATIONS:
Overall Officials: John Kane, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States